CLINICAL TRIAL: NCT00243438
Title: Distinctly Access Vision In Coronary Interventions
Brief Title: DaVinci Registry(Distinctly Assess Vision in Coronary Intervention)
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Matt Kiely, Abbott Vascular
Other Study IDs: Version vom 18.7.2003
Record Dates: First submitted 2005-10-21; First posted 2005-10-24 (Estimated); Last update posted 2009-01-28 (Estimated); Status verified 2009-01

CONDITIONS: Coronary Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Patients who have received a Vision stent and who have diabetes and/or complex lesions.
  Interventions: Device: Multilink Vision™ Stent (CE-labeled)

INTERVENTIONS:
Device: Multilink Vision™ Stent (CE-labeled) — Patients who have diabetes and/or complex lesions and who have had a Multilink Vision™ Stent placed.

SUMMARY:
Prospective Internet-Registry, Postmarketing-Surveillance, Registration and Follow-up of patients after Multi-Link VISION™ - Stent Implantation

DETAILED DESCRIPTION:
A Non-Randomized prospective evaluation of the Multi-Link Rx Vision TM Coronary Stent System in the treatment of patients with De novo native coronary artery lesions

ELIGIBILITY:
Inclusion Criteria:

* Women and Men Age >18 years, Intention to treat all stenosis with Multi-Link VisionTM Stents, documented patient consent

Exclusion Criteria:

* No Multi-Link Vision™ Stent implanted, life expectation >9 M, cardiogenic shock, STEMI, NSTEMI or unstable angina pectoris with pathologic markers within the last 48 hours, intolerance of Clopidogrel/ Tiklopidin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diabetes and/or complex coronary artery disease who are treated with a Multi-Link Vision™ Stent.
Sampling Method: Non-Probability Sample
Enrollment: 1300
Dates: Start 2003-07; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
TVF | 9 months

SECONDARY OUTCOMES:
Mode of death
Time to first MI
TVR
CABG

CONTACTS AND LOCATIONS:
Overall Officials: Christian Hamm, MD, Principal Investigator — Kerckhoff-Klinik/ Benekestr. 2-8/ 61231 Bad Nauheim
Locations (1):
- Kerckhoff-Klinik, Bad Nauheim, Germany